CLINICAL TRIAL: NCT06821737
Title: Diagnostic Accuracy of Using Point-of-care Ultrasonography for Confirming Nasogastric Tube Placement: a Multicentre Prospective Study
Brief Title: Diagnostic Accuracy of Using Point-of-care Ultrasonography for Confirming Nasogastric Tube Placement
Status: Active, not recruiting | Type: Observational
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Mak Mei Yi, Nurse Consultant, Pamela Youde Nethersole Eastern Hospital
Other Study IDs: CIRB-2024-467-2
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Ultrasound; Nasogastric Tube; Nasogastric Tube Placement
MeSH Terms: interventions — Ultrasonography; Radiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Observational Group: All participants included will be in one observational cohort.
  Interventions: Device: Diagnostic ultrasound; Device: Diagnostic X-ray

INTERVENTIONS:
Device: Diagnostic ultrasound — A portable wireless ultrasound system (Vscan Air, General Electric Healthcare) with dual probes-linear array (3-12 MHz) for neck scanning and curved array (2-5 MHz) for subxiphoid scanning-will be used. The linear probe is placed transversely on the anterior neck, slid left at the thyroid level to focus on the esophagus, then rotated for longitudinal views. The curved probe is applied subxiphoid, using the liver as a landmark, and tilted left to image the stomach. A positive result is confirmed by visualizing the NGT shadow in the esophagus and stomach, followed by dynamic upsurge fogging after injecting 50cc of air. Ultrasonography and X-ray results will be compared.
Device: Diagnostic X-ray — This study will employ chest radiography as the reference standard for verification of correct nasogastric tube placement. Radiographic imaging will be conducted following NGT insertion and interpreted by physicians to verify positional accuracy.

SUMMARY:
A prospective observational diagnostic study will be conducted to assess the sensitivity and specificity of ultrasound in verifying the correct nasogastric tube placement, using X-ray as the reference standard.

DETAILED DESCRIPTION:
This study is a prospective observational diagnostic investigation aimed at evaluating the accuracy of ultrasound in confirming nasogastric tube (NGT) placement. Participants aged 18 years or older requiring NGT insertion will be recruited via convenience sampling from community nursing centres across five clusters and medical and geriatric wards in four acute or convalescent hospitals. Nurses performing index tests will complete standardized POCUS training (8-hour theory and practical sessions, written exams, 3-month bedside practicum with ≥20 positive scans) prior to competency assessment. Direct visualisation of an NGT in both the oesophagus and stomach will be interpreted as correct stomach placement. When the acoustic shadow of an NGT was not seen in the stomach, 50cc of air was injected through the NGT, and it was considered well-placed if the ultrasonography showed dynamic fogging. Correct gastric placement is assumed if the acoustic shadow of an NGT is visible in the oesophagus and stomach, even if fogging is not detectable. The reference standard will be post-index test X-ray confirmation. Diagnostic performance metrics, including sensitivity, specificity, positive and negative predictive values, and likelihood ratios, will be calculated to assess the efficacy of ultrasound. Variability in diagnostic accuracy across participant characteristics will be analyzed. Additionally, the study will compare the time intervals between ultrasound and X-ray, delays in feeding initiation post-placement, and associated costs, including emergency department admissions, unplanned hospitalizations, and ambulance transportation.

The findings will provide critical evidence on the diagnostic utility of ultrasound for NGT placement verification, informing potential revisions to clinical practice guidelines and supporting stakeholder decisions on integrating ultrasound as a reference test.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older;
* Living in the community or admitted to a medical and geriatric ward;
* Requiring the use of an NGT during the recruitment period for assessment, monitoring, nutritional assistance, drainage, and/or medication administration;
* Aspirated fluids with a pH value of more than 5.5 after insertion or with insufficient fluids for pH testing after insertion;

Exclusion Criteria:

* Uncooperative patients;
* Had head and neck injury
* Have had a gastrectomy or by-pass surgery;
* History of abdominal trauma or receiving emergency life support intervention at time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience sampling will be adopted in this study. Participants will be recruited from six community nursing centres in Hong Kong East, Hong Kong West, Kowloon Central, Kowloon West, and New Territories West Cluster hospitals, as well as 38 wards from medical and geriatric wards across 4 acute, rehabilitation or convalescent hospitals managed by the Hospital Authority. Participants will be engaged by episodes throughout the study.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Ultrasound in correct Nasogastric Tube placement confirmation | An average of 18 months
  Sensitivity: True Positive / (True Positive + False Negative) x 100% Specificity: True Negative / (True Negative + False Positive) x 100% Positive Predictive Value: True Positive / (True Positive + False Positive) x 100% Negative Predictive Value: True Negative / (True Negative + False Negative) x 100% Positive Likelihood Ratio: sensitivity / 1 - specificity Negative Likelihood Ratio: 1 - sensitivity / specificity

SECONDARY OUTCOMES:
Time lag between USG & x-ray | An average of 18 months
  The study will assess the time lag between ultrasound confirmation and subsequent X-ray imaging for nasogastric tube placement verification.
Delay between tube placement and feeding by x-ray | An average of 18 months
  The study will evaluate the delay between nasogastric tube placement and the initiation of feeding, as confirmed by X-ray.
Cost of ED admission, unplanned admission, ambulance transportation | An average of 18 months
  The study will analyze costs associated with Emergency Department admissions, unplanned hospital admissions, and ambulance transportation related to nasogastric tube placement confirmation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Authority, HKSAR, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during this study will be made available by the principal investigator upon reasonable request.

REFERENCES:
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig L, Lijmer JG, Moher D, Rennie D, de Vet HC, Kressel HY, Rifai N, Golub RM, Altman DG, Hooft L, Korevaar DA, Cohen JF; STARD Group. STARD 2015: an updated list of essential items for reporting diagnostic accuracy studies. BMJ. 2015 Oct 28;351:h5527. doi: 10.1136/bmj.h5527. PMID 26511519
- [Background] Zatelli M, Vezzali N. 4-Point ultrasonography to confirm the correct position of the nasogastric tube in 114 critically ill patients. J Ultrasound. 2016 Oct 28;20(1):53-58. doi: 10.1007/s40477-016-0219-0. eCollection 2017 Mar. PMID 28298944
- [Background] Wong KW, Chan HH, Wong CP, Chan MY, Chau JCW, Wong TW. Using color flow detection of air insufflation to improve accuracy in verifying nasogastric tube position. Am J Emerg Med. 2017 Feb;35(2):333-336. doi: 10.1016/j.ajem.2016.12.046. Epub 2016 Dec 21. PMID 28038826
- [Background] Tsujimoto Y, Kataoka Y, Banno M, Anan K, Shiroshita A, Jujo S. Ultrasonography for confirmation of gastric tube placement. Cochrane Database Syst Rev. 2024 Jul 25;7(7):CD012083. doi: 10.1002/14651858.CD012083.pub3. PMID 39051488
- [Background] Nedel WL, Jost MNF, Filho JWF. A simple and fast ultrasonographic method of detecting enteral feeding tube placement in mechanically ventilated, critically ill patients. J Intensive Care. 2017 Aug 18;5:55. doi: 10.1186/s40560-017-0249-5. eCollection 2017. PMID 28828174
- [Background] Mumoli N, Vitale J, Pagnamenta A, Mastroiacovo D, Cei M, Pomero F, Giorgi-Pierfranceschi M, Giuntini L, Porta C, Capra R, Mazzone A, Dentali F. Bedside Abdominal Ultrasound in Evaluating Nasogastric Tube Placement: A Multicenter, Prospective, Cohort Study. Chest. 2021 Jun;159(6):2366-2372. doi: 10.1016/j.chest.2021.01.058. Epub 2021 Feb 2. PMID 33545162
- [Background] McMullen CD, Anstey C, Garrett P, Moore J. Nasogastric tube placement under sonographic observation: A comparison study of ultrasound and chest radiography in mechanically ventilated patients. Aust Crit Care. 2022 Mar;35(2):181-185. doi: 10.1016/j.aucc.2021.03.006. Epub 2021 Jun 11. PMID 34120804
- [Background] Mak MY, Tam G. Ultrasonography for nasogastric tube placement verification: an additional reference. Br J Community Nurs. 2020 Jul 2;25(7):328-334. doi: 10.12968/bjcn.2020.25.7.328. PMID 32614666
- [Background] Lin T, Gifford W, Lan Y, Qin X, Liu X, Wang J, Yang B, You T, Chen K. Diagnostic accuracy of ultrasonography for detecting nasogastric tube (NGT) placement in adults: A systematic review and meta analysis. Int J Nurs Stud. 2017 Jun;71:80-88. doi: 10.1016/j.ijnurstu.2017.03.005. Epub 2017 Mar 9. PMID 28359986
- [Background] Gok F, Kilicaslan A, Yosunkaya A. Ultrasound-guided nasogastric feeding tube placement in critical care patients. Nutr Clin Pract. 2015 Apr;30(2):257-60. doi: 10.1177/0884533614567714. Epub 2015 Jan 23. PMID 25616518
- [Background] Brun PM, Chenaitia H, Lablanche C, Pradel AL, Deniel C, Bessereau J, Melaine R. 2-point ultrasonography to confirm correct position of the gastric tube in prehospital setting. Mil Med. 2014 Sep;179(9):959-63. doi: 10.7205/MILMED-D-14-00044. PMID 25181712